CLINICAL TRIAL: NCT00722033
Title: Effect of Common Neonatal Procedures Over the Amplitude- Integrated Electroencephalography Register in <30 Weeks Preterms.
Brief Title: Common Neonatal Procedures Could Affect the aEEG in <30 Weeks of Gestational Age Preterms
Acronym: ELECTROPREM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Paulina Toso/MD, Pontificia Universidad Catolica
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PontificiauCC
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-07

CONDITIONS: Regional Blood Flow; Premature Birth; Electroencephalography
Keywords: preterm; aEEG; apneas; surfactant; indomethacin; aminophyline
MeSH Terms: conditions — Premature Birth; Apnea | interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): < 30 weeks of gestation
  Interventions: Drug: 3 protocols of Indomethacin administration

INTERVENTIONS:
Drug: 3 protocols of Indomethacin administration — Indomethacin will consecutive be infused in 30, 60 and 120 minutes in each patient who requires it.
  Other Names: indomethacin

SUMMARY:
Very low birth weight infants has increased dramatically their survival. Survival without neurologic disturbance varies a lot between centers.There is evidence that fluctuations in cerebral blood flow influences the appearance of intraventricular hemorrhage and itself implies a detrimental neurologic developing.The electroencephalography is the result of electric base membrane activity on rest, and it's influenced by the blood flow either. The Amplitude-integrated electroencephalography is a novel tool, that is capable to be continuously used at the patient bed and is easily to be read by the trained clinician.The hypothesis is that common procedures as Surfactant instilation, Indomethacin and Aminophyline infusion as the appearance of apneas alters the aEEG register. It is a prospective study that tries to recruit 10 < 30 weeks of gestational age with aprofen consent to monitorize the aEEG since birth to the seventh day of live.

DETAILED DESCRIPTION:
The survival of extreme premature babies ( < 1000 grams) has improved in the last years. The neonatal networks have realized of these results and of the interventions associated with better forecast in the managing of certain punctual problems. Also they have informed that differences exist in the results obtained among the centers credited for the managing of this type of patients. One of the challenges of the current Neonatology is the survival without sequels.

It is of principal worry the neurological sequels in the extreme premature babies. These can go from severe alterations up to minimal disorders. The managing of the critical patient includes the strict and continuous monitoring of the vital signs. The cerebral function is of evaluation limited in the acute period of these patients. The electroencephalography is the expression of the membrane potential in rest neuronal. One has seen that the changes in cerebral flow affect the electrical sign emitted by this one. There have been reported that some conditions that in the neonatal period are associated with alterations of cerebral flow. This way there is described, that the application of surfactant is associated with fluctuations of the cerebral flow, the arterial unbalanced ductus, Indomethacin's injection in less than 30 minutes, episodes of severe hypoxemia , Methylxanthines's injection,etc.

For some years there is used the Monitoring of Amplitude-Integrated Electroencephalography to term newborn.It corresponds to the Electroencephalography sign obtained in C3 and C4 location of the standard electroencephalography, amplification of the sign, filtered to 2-15Hz, submitted to a semilogarithmic compression of the extent rectified by a constant of time of 0,5 seconds and compressed. This gives origin to different patterns, possible to interpret for the clinician in real time. The use of this tool in premature babies is still experimental.

It is tried to evaluate if common procedures theorically associated with alteration of the cerebral flow, in extreme premature babies affect the Amplitude- Integrated Electroencephalography record. It will measure up if changes happen to relation to the application of Surfactant, Indomethacin in 3 rate of application and Aminophyline's infusion. The effect of desaturation will measure up, bradycardias and apneas in the extent of voltage.

For this they will be monitored in continuous form from the birth to 10 premature babies <30 weeks of gestational age for 7 days, previous obtaining of informed consent. Protocols will be applied:quality of sign and specifics according to the raised aims. The analysis will be done by means of programs EEG Viewer and Chart Analyzer.The analysis of the bosses of aEEG and of his variations will be realized manually, applying the Burdjalov and Spitzer score. The periods before, during and after the administration of Surfactant, Indomethacin and Aminophyline were selected . In case of apneas, bradycardias and desaturation it will be compared 1 minute before with the properly such episode. These episodes will be transfer to an Excel schedule for his numerical analysis. This will allow the obtaining of averages and standard diversion of the extent of voltage of every episode and it's going to be calculated if there is any difference before and after each episode. The same is going to be done for Surfactant (5 minutes before and after), Indometacin(30 minutes before and during the 3 rates of infusion) and Aminophyline(15 minutes before and after) The level of statistics significance for all the test will be p < 0,05.

One expects to achieve ideal quality of sign > 75 % of the registered time. One tries to evaluate 12 Surfactant applications, 35 of Indomethacin, 60 of Aminophyline and 100 cardiorespiratory events. One expects to find differences in the Extent of voltage in relation to desaturations, bradycardias and apneas.

ELIGIBILITY:
Inclusion Criteria:

* < 30 weeks of gestational age
* Consent inform approved

Exclusion Criteria:

* Known mayor malformation

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
aEEG voltage amplitude changes after procedures | right after procedure

SECONDARY OUTCOMES:
aEEG amplitude voltage changes between 3 administration protocols of Indomethacin | right after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Puc, Nicu, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Burdjalov VF, Baumgart S, Spitzer AR. Cerebral function monitoring: a new scoring system for the evaluation of brain maturation in neonates. Pediatrics. 2003 Oct;112(4):855-61. doi: 10.1542/peds.112.4.855. PMID 14523177
- [Background] Hellstrom-Westas L, Rosen I. Continuous brain-function monitoring: state of the art in clinical practice. Semin Fetal Neonatal Med. 2006 Dec;11(6):503-11. doi: 10.1016/j.siny.2006.07.011. Epub 2006 Oct 24. PMID 17067863